CLINICAL TRIAL: NCT05444621
Title: Carotid Ultrasounds Measurements for Assessment of Fluid Responsiveness in Septic Shock
Brief Title: Carotid Ultrasounds Measurements in Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Abdelhameed Mohammed Hassan, principal investigator, Assiut University
Other Study IDs: carotid US
Record Dates: First submitted 2022-06-20; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Ultrasound and doppler — All patients are then assessed by transthoracic echocardiography to measure Left ventricle and Right ventricle function and to assess LVOT-VTI and SV. Doppler Ultrasound assessment of carotid arteries to assess corrected flow time (FTc), velocity time integral (VTI) and respirophasic variation in carotid artery blood flow peak velocity (ΔVpeak). The patient will be assessed pre- and post- passive leg raising (PLR) and after fluid challenge of 30 mL/Kg of IV crystalloid

SUMMARY:
The aim of the study is to assess carotid ultrasounds measurements, namely corrected flow time (FTc), velocity time integral (VTI) and respirophasic variation in carotid artery blood flow peak velocity (ΔVpeak), as a predictor of fluid responsiveness in septic shock patients.

DETAILED DESCRIPTION:
Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection . Early identification and appropriate management in the initial hours after the development of sepsis improve outcomes.

For patients with sepsis-induced hypoperfusion or septic shock it is recommended to give IV crystalloid fluid within the first 3 hr of resuscitation . However, fluid responsiveness varies widely between cases. Determining the optimal amount of fluid to be administered remains a critical issue in clinical practice and research. Recent studies have shown that not every patient advantages from intravenous hydration, only 40% of hypotensive patients with sepsis benefit, and the others who do not respond are liable to develop pulmonary edema with high associated mortality . Studies have shown that aortic blood peak velocity had high sensitivity and specificity to predict fluid responsiveness, however, measurements of aortic blood flow velocity need a transesophageal ultrasound which is an invasive procedure . Measurement of left ventricular outflow tract velocity time integral (LVOTVTI), derived stroke volume (SV), and cardiac output reliably predicts fluid responsiveness in critically ill patients but it is difficult and dependent on operator and echo windows . There is a need to find a non-invasive accurate and easy method to assess fluid responsiveness in septic shock patients. Different Measurements of carotid artery flow have been suggested recently to predict fluid responsiveness. A promising measurements are corrected flow time (FTc), velocity time integral (VTI) and respirophasic variation in carotid artery blood flow peak velocity (ΔVpeak).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 year old) diagnosed with septic shock (MAP >65mmHg), within 6 hours of admission or development of septic shock if previously admitted with other diagnoses.

Exclusion Criteria:

* patients have any of these conditions: Carotid artery stenosis ≥50%, known heart failure (Ejection fraction ≤45%) or End Stage Kidney Disease requiring haemodialysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All recruited patients aged between 18 and 75 year old suspected to have septsis and septic shock are to be assessed at time of admission by history taking, thorough physical examination, laboratory workup. ECG, haemodynamic parameters and abdominal ultrasound including inferior vena cava (IVC) dimeter and collapsibility. Sequential Organ failure Assessment (SOFA) and Acute Physiology and Chronic Health Evaluation (APACHE-II) score to diagnose septic shock and eligibility to enter the study .
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
carotid usltrasounds and doppler measurements as predictor of fluid responsiveness in septic patient | baseline
  Assess carotid artery blood flow assessed by Ultrasounds as a predictor of fluid responsiveness in septic shock patients, and compare this measurements to standard one as echocardiography measurements of stroke volume and cardiac output (COP)to establish more easier method for assessment not depend of echo-window of patient and doesn't need expert one to do.

REFERENCES:
- See also: Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. — https://link.springer.com/article/10.1007/s00134-021-06506-y?fbclid=IwAR022PGaW_CAvqLEy7QL3sW_JTa_QqG0cEjeWHljJrVqm_aGf18BkCfs9F4
- See also: Wu Y, Zhou S, Zhou Z, Liu B. A 10-second fluid challenge guided by transthoracic echocardiography can predict fluid responsiveness. Crit Care. 2014;;18::R108.. doi: 10.1186/cc13891. DOI: — https://ccforum.biomedcentral.com/articles/10.1186/cc13891
- See also: Sidor M, Premachandra L, Hanna B, Nair N, Misra A. Carotid flow as a surrogate for cardiac output measurement in Hemodynamically stable participants. J Intensive Care Med. 2020;;35::650--655.. doi: 10.1177/0885066618775694. DOI: — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7991757/